CLINICAL TRIAL: NCT05048667
Title: Novel Treatment for Microvascular Erectile Dysfunction Combining Shockwave Therapy and Platelet Rich Plasma
Brief Title: Shockwave Therapy and Platelet Rich Plasma for the Treatment of Erectile Dysfunction
Acronym: COCKTAIL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Emad Ibrahim, Assistant Professor of Clinical Urology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20210887; R01DK130991 (NIH)
Record Dates: First submitted 2021-09-07; First posted 2021-09-17 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- SWT plus PRP Group (Experimental): Participants will receive weekly Shockwave Therapy (SWT) and Platelet Rich Plasma (PRP) for 5 weeks. SWT will be administered weekly on Weeks 1, 2, 3, 4, and 5. PRP will be administered on Week 1 and Week 5.
  Interventions: Device: Shock Wave therapy (SWT); Drug: Platelet Rich Plasma (PRP)
- Sham SWT plus Placebo Saline Group (Placebo Comparator): Participants will receive weekly Sham Shockwave Therapy (SWT) and Placebo Saline Intracavernosal Injection (ICI) for 5 weeks. Sham SWT will be administered weekly on Weeks 1, 2, 3, 4, and 5. Placebo Saline ICI will be administered on Week 1 and Week 5.
  Interventions: Other: Sham SWT; Other: Placebo Saline

INTERVENTIONS:
Device: Shock Wave therapy (SWT) — Each SWT will administer 720 shocks in the treatment arm. Total of 3600 shocks are given over 5 weeks treatment period.
  Arms: SWT plus PRP Group
Drug: Platelet Rich Plasma (PRP) — 5 mL PRP will be administered via intracavernous injection
  Arms: SWT plus PRP Group
Other: Sham SWT — Sham Shockwave Therapy will be administered in the sham arm.
  Arms: Sham SWT plus Placebo Saline Group
Other: Placebo Saline — 5 mL Placebo saline will be administered via intracavernous injection in the sham arm.
  Arms: Sham SWT plus Placebo Saline Group

SUMMARY:
The purpose of this research study is to evaluate whether the combination of Shock Wave Therapy (SWT) with Platelet Rich Plasma (PRP) is synergistic and can reverse the pathology of microvascular Erectile Dysfunction (ED) and enhance erectile function by improving vasodilation, and endothelial function

ELIGIBILITY:
Inclusion Criteria:

1. Be Male
2. Be 30 to 80 years of age (inclusive).
3. Be able to provide written informed consent.
4. Have a diagnosis of ED due to organic origin for at least 6 months prior to consent.
5. Sexually active in a stable, heterosexual relationship of more than three months duration.
6. IIEF-EF score 12-25 at screening
7. Agree to attempt sexual intercourse at least 4 times per month for the duration of the study without being under the influence of alcohol or recreational drugs.
8. Agree to comply with all study related tests/procedures.

Exclusion Criteria:

1. Previous penile surgery of any kind (except circumcision and condyloma removal), such as penile lengthening, penile cancer surgery, penile plication, grafting.
2. Previous history of priapism or penile fracture
3. Abnormal morning serum testosterone level defined as a value lower than 300 ng/dL (±5%) (indicative of untreated hypogonadism), or greater than 1197 ng/dL (±5%).
4. Current or previous hormone usage, other than prescribed testosterone, clomiphene or thyroid medication. (Subjects with prior or current use of hormonal treatment for prostate cancer are also excluded.
5. Psychogenic ED as determined by study investigator.
6. Anatomical (Peyronie's Disease or penile curvature that negatively influences sexual activity) or neurological abnormalities in the treatment area.
7. Patients using Intracavernosal Injection (ICI) for management of ED
8. Patients with generalized polyneuropathy, or neurological conditions irrespective of cause, such as severe diabetes, multiple sclerosis or Parkinson's disease.
9. Have a serious comorbid illness/condition/behavior that, in the opinion of the investigator, may compromise the safety or compliance of the subject or preclude successful completion of the study.
10. History of consistent treatment failure with Phosphodiesterase Type 5 (PDE5) inhibitors for therapy of ED.
11. Any history of significant psychiatric disease, such as bipolar disorder or psychosis, greater than one lifetime episode of major depression, current depression of moderate or greater severity. Patients who are currently using Selective Serotonin Reuptake Inhibitors (SSRI) or psychotropic medications.
12. Hemoglobin a1c >9%.

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Change in IIEF-EF Scores | Baseline, Month 3, Month 6
  International Index of Erectile Function - Erectile Function Subdomain Score (IIEF-EF) is a 5-item subdomain self- evaluation questionnaire of erectile function with a total score ranging from 0-25 with the higher score indicating better erectile function.
Percentage of participants achieving MCID in IIEF-EF | Baseline, Month 3, Month 6
  IIEF-EF is a 5-item subdomain self- evaluation questionnaire of erectile function with a total score ranging from 0-25 with the higher score indicating better erectile function. Mild Clinically Important Difference (MCID) is attained via an increase of 2 points in IIEF-EF score for participants with mild ED and an increase of 5 points for participants with moderate ED.
Penile Blood Flow | Baseline, Month 6
  Penile Blood Flow will be reported as Peak Systolic Velocity (PSV) and End Diastolic Velocity (EDV), both assessed in cm/sec, via Penile Doppler ultrasonography
Circulating Angiogenic Factor levels | Baseline, Month 3, Month 6
  Circulating angiogenic factor levels including Vascular Endothelial Growth Factor (VEGF), Stromal Cell Derived Factor-1 (SDF-1 alpha) and Stem cell Factor (SCF), all reported in pg/mL, will be assessed via blood samples

SECONDARY OUTCOMES:
Number of participants reporting a decrease or discontinue in use of PDE5 inhibitors | Baseline, Month 3
  The number of participants reporting a decrease or discontinue in use of PDE5 inhibitors will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Emad Ibrahim, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Miller School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andia I, Maffulli N. Platelet-rich plasma for managing pain and inflammation in osteoarthritis. Nat Rev Rheumatol. 2013 Dec;9(12):721-30. doi: 10.1038/nrrheum.2013.141. Epub 2013 Oct 1. PMID 24080861
- [Background] Sampson S, Gerhardt M, Mandelbaum B. Platelet rich plasma injection grafts for musculoskeletal injuries: a review. Curr Rev Musculoskelet Med. 2008 Dec;1(3-4):165-74. doi: 10.1007/s12178-008-9032-5. PMID 19468902
- [Background] Xie X, Zhang C, Tuan RS. Biology of platelet-rich plasma and its clinical application in cartilage repair. Arthritis Res Ther. 2014 Feb 25;16(1):204. doi: 10.1186/ar4493. PMID 25164150
- [Background] Randelli P, Randelli F, Ragone V, Menon A, D'Ambrosi R, Cucchi D, Cabitza P, Banfi G. Regenerative medicine in rotator cuff injuries. Biomed Res Int. 2014;2014:129515. doi: 10.1155/2014/129515. Epub 2014 Aug 13. PMID 25184132
- [Background] Vlachopoulos C, Rokkas K, Ioakeimidis N, Aggeli C, Michaelides A, Roussakis G, Fassoulakis C, Askitis A, Stefanadis C. Prevalence of asymptomatic coronary artery disease in men with vasculogenic erectile dysfunction: a prospective angiographic study. Eur Urol. 2005 Dec;48(6):996-1002; discussion 1002-3. doi: 10.1016/j.eururo.2005.08.002. Epub 2005 Aug 24. PMID 16174548
- [Background] Haupt G, Haupt A, Ekkernkamp A, Gerety B, Chvapil M. Influence of shock waves on fracture healing. Urology. 1992 Jun;39(6):529-32. doi: 10.1016/0090-4295(92)90009-l. PMID 1615601
- [Background] Melman A, Gingell JC. The epidemiology and pathophysiology of erectile dysfunction. J Urol. 1999 Jan;161(1):5-11. PMID 10037356
- [Background] Kikuchi Y, Ito K, Ito Y, Shiroto T, Tsuburaya R, Aizawa K, Hao K, Fukumoto Y, Takahashi J, Takeda M, Nakayama M, Yasuda S, Kuriyama S, Tsuji I, Shimokawa H. Double-blind and placebo-controlled study of the effectiveness and safety of extracorporeal cardiac shock wave therapy for severe angina pectoris. Circ J. 2010 Mar;74(3):589-91. doi: 10.1253/circj.cj-09-1028. Epub 2010 Feb 4. PMID 20134096
- [Derived] Saltzman RG, Molina ML, Ledesma BR, Ibrahim E, Masterson TA, Ramasamy R. Rationale and Design for the COCKTAIL Trial: A Single-center, Randomized, Double-blind, Sham-controlled Study Combining Shockwave Therapy and Platelet-rich Plasma for Erectile Dysfunction. Eur Urol Focus. 2023 Jan;9(1):8-10. doi: 10.1016/j.euf.2022.09.015. Epub 2022 Oct 22. PMID 36280578